CLINICAL TRIAL: NCT06755554
Title: Investigation of Effect of Indocyanine Green on Volume of Lymph Node Dissection in Surgical Treatment of Gastric Cancer
Brief Title: Investigation of Impact of Indocyanine Green on Volume of Lymphadenectomy in Resectable Gastric Cancer
Acronym: ICGastr
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ukrainian Society of Clinical Oncology (Other)
Responsible Party: Principal Investigator, Oleksii Dobrzhanskiy, Doctor, Ukrainian Society of Clinical Oncology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 272/4
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Gastric Cancer Stage II; Gastric Cancer Stage III; Gastric Cancer; Gastrectomy for Gastric Cancer
Keywords: indocyanine green; gastric cancer; gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Indocyanine green mapping (Experimental): Endoscopic injection of indocyanine green is performed under general anesthesia.
  Indocyanine green is injected into the submucosal layer of the stomach at 4 points around the tumor. The dosage for one administration is up to 5 mg. The total dosage for one patient for 4 doses is 20 mg. Monitoring of indocyanine green side effects occurs before the start of general anesthesia during radical surgery.
  Interventions: Drug: Endoscopic injection of Indocyanine green

INTERVENTIONS:
Drug: Endoscopic injection of Indocyanine green — ICG is injected by the patient by endoscopic submucosal injection into 4 points around the tumor 24-12 hours before the start of the surgical intervention.

SUMMARY:
The study aims to evaluate the safety and benefits of using indocyanine green in lymph node dissection for gastric cancer surgery. The primary endpoint is the average number of lymph nodes removed. Secondary study points are the average number of ICG-positive lymph nodes; the average number of metastatic ICG-positive lymph nodes; the number of postoperative complications and complications associated with the administration of ICG.

Patients who meet the inclusion criteria for this study will be enrolled in the study after reviewing and signing an informed consent form.

All patients will be included in one group and will receive surgical treatment in the amount of total or subtotal gastrectomy with lymphadenectomy D1, D1+, D2 or D2+.

ICG is injected by the patient by endoscopic submucosal injection into 4 points around the tumor 24-12 hours before the start of the surgical intervention.

Assessment of the number of fluorescent lymph nodes will be performed intraoperatively with their subsequent removal and mapping. The incidence of postoperative complications will be assessed by Clavien-Dindo.

DETAILED DESCRIPTION:
1. Introduction and rationale Radical gastrectomy with D2 lymph node dissection remains the main treatment for resectable gastric adenocarcinoma. Lymph node status is a significant prognostic factor for the survival of patients with gastric cancer, as high-quality lymph node dissection improves patient prognosis. However, lymph node dissection in gastric cancer surgery is sometimes not performed in full and is routinely performed without the use of additional imaging methods. As a result, a complete lymphadenectomy is technically difficult, which leads to smaller lymphadenectomies and, in turn, to tumor recurrence and poorer overall survival rates for this group of patients. The use of intraoperative navigation technology to assist in systemic lymph node dissection is essential for radical gastrectomy.

   The sentinel lymph node (SLN) is defined as the first lymph node on the path of lymphatic drainage from the primary tumor. Currently, the method of labeling the SLN is widely used in the treatment of tumors of various localizations. Gastric cancer has also been identified as an object for signal node navigation surgery. The results of studies indicate that sentinel lymph node navigation surgery can become the basis for minimally invasive surgery with personalized lymphadenectomy and improve the treatment outcomes and quality of life of patients with various types of malignancies, including gastric cancer.

   Dyes, radioisotopes, or a combination of both are used to label SLNs in gastric cancer. However, they all have certain limitations that make it impossible to use them routinely.

   Indocyanine green (ICG) is a well-known diagnostic reagent that is approved for clinical use in the study of liver function and cardiac output. It absorbs light in the near-infrared with a maximum at 800 nm and emits maximum fluorescence at 840 nm when bound to plasma proteins. Based on the fluorescence characteristics of IR, an intraoperative imaging system was developed to assess blood flow during surgical interventions, such as coronary artery bypass grafting, neurovascular surgery, and organ transplantation. In addition, the use of fluorescence imaging has been widely used for labeling of SLAs in cancer.
2. The purpose of the study The study aims to evaluate the safety and benefits of using indocyanine green in lymph node dissection for gastric cancer surgery. The primary endpoint is the average number of lymph nodes removed. Secondary study points are the average number of ICG-positive lymph nodes; the average number of metastatic ICG-positive lymph nodes; the number of postoperative complications and complications associated with the administration of ICG.
3. Design. This study is a prospective, open-label, single-center clinical trial with one study group to investigate the number of lymph nodes removed using ICG.

   Patients who meet the inclusion criteria for this study will be enrolled in the study after reviewing and signing an informed consent form.

   All patients will be included in one group and will receive surgical treatment in the amount of total or subtotal gastrectomy with lymphadenectomy D1, D1+, D2 or D2+.

   ICG is injected by the patient by endoscopic submucosal injection into 4 points around the tumor 24-12 hours before the start of the surgical intervention.

   Assessment of the number of fluorescent lymph nodes will be performed intraoperatively with their subsequent removal and mapping. The incidence of postoperative complications will be assessed by Clavien-Dindo.
4. Study population 4.1 General data The study population consists of patients with newly diagnosed gastric cancer of stages Ib, II, III. Patients are treated according to national standards for the treatment of gastric cancer.

   4.2 Inclusion criteria: A. Tumor spread: cT2-4a cN0-3, cM0; B. Age: 18 - 80; C. Gender: men and women; D. ECOG: 0 - 1; E. Histologic type of tumor: Adenocarcinoma of any subtype; F. Degree of differentiation: G1 - G4; G. Tumor localization: cardiac region, stomach floor, stomach body, antrum, pylorus, and pyloric region of the stomach; H. Tumor spread: absence of tumor invasion into adjacent structures; I. No history of cancer in the last 5 years. J. No previous chemotherapy, surgery or radiation treatment for another cancer (except for neoadjuvant chemotherapy for gastric cancer); K. Absence of decompensated concomitant pathology.

   4.3. Exclusion criteria : A. M1 (distant metastases); B. ECOG 2 - 4; C. Age over 80 and under 18; D. Presence of decompensated comorbidities, ASA> 3; E. Patient refusal to participate in the study.
5. Statistics 5.1 Sample calculation According to the literature, the average number of lymph nodes removed is 48.9 (+- 14.6). An increase in the average number of lymph nodes by 4 will be sufficient to reject the null hypothesis with 80% power and a one-sided significance criterion of 0.05. This will require the recruitment of 105 patients. Patient recruitment is planned over a three-year period, with each patient followed for 90 days after surgical treatment. About 30 patients are planned to be included each year.

   5.2 Analysis. The primary endpoint analysis is planned in accordance with the intention-to-treat provision, which provides for the analysis of all patients who will be included in the study, regardless of the treatment and its effect.

   The difference in the mean number of lymph nodes will be analyzed using the t-test. For the analysis of other treatment-related complications, multivariate analysis will be used for each clinical factor and its association with the development of the main types of complications. Continuous data will be analyzed using the unpaired Student's t-test. Multivariate analysis to determine the correlation between clinical variables and complications will be performed using a logistic regression model.
6. Quality control 6.1 Quality criteria for surgical intervention

   The criterion for the quality of indocyanine green injection will be intraoperative visual assessment of lymph node fluorescence, visual assessment of adjacent tissue fluorescence. The quality of lymph node dissection will be assessed by the number of lymph nodes removed and the number of lymph node groups removed for each patient and the R-status of the lymph nodes (R0/R1/R2). The quality of gastric tumor removal will be assessed by evaluating the resection margins (R0/R1/R2).

   6.2 Protocol for recording complications associated with indocyanine administration and postoperative complications The frequency and nature of complications associated with the administration of indocyanine green will be assessed according to the Common Terminology Criteria for Adverse Events 5.0. The frequency and nature of surgical complications will be assessed according to the Clavien-Dindo classification.
7. Algorithm of patient registration and inclusion in the study After signing the informed consent, a unique number will be assigned to the patient, which will be entered into the paper CRF form and duplicated in the electronic . The paper form and the electronic database completely duplicate each other. The electronic form and the paper form are filled in by the researcher as soon as the patient signs the informed consent to participate in the study. The electronic form is based on the Redcap database.

8.1 Principles of administration of green indocyanine Before endoscopic injection of indocyanine green and surgical treatment, the tests listed in Appendix 6 are required.

Endoscopic injection of indocyanine green is performed under general anesthesia.

Indocyanine green is injected into the submucosal layer of the stomach at 4 points around the tumor. The dosage for one administration is up to 5 mg. The total dosage for one patient for 4 doses is 20 mg. Monitoring of indocyanine green side effects occurs before the start of general anesthesia during radical surgery.

8.2 Principles of clinical and laboratory monitoring Clinical and laboratory monitoring of patients is performed before the administration of indocyanine green and the start of surgery. If side effects occur between the administration of indocyanine green and the beginning of general anesthesia for carrying out curative surgery, it is possible to conduct additional clinical and laboratory examinations at the discretion of the investigator.

8.3 List of tests for the administration indocyanine green and radical surgical treatment See Annex 6.

8.4 Principles of surgical treatment Surgical treatment of gastric cancer is performed in accordance with national guidelines for the treatment of gastric cancer. The main goal of surgery is: radical removal of the tumor; achievement of R0 status of the resection margins; lymph node dissection in the volume corresponding to the volume of the primary tumor removal (D1/D1+/D2/D2+).

Criteria for gastric cancer unresectability:

● invasion of the following vessels: aorta, vena cava, abdominal trunk, common hepatic artery, hepatic artery proper, left hepatic artery, right hepatic artery, portal vein, liver parenchyma.

9. Postoperative patient management. In 16-20 hours after the end of the surgery, the patient starts drinking water (50 ml per dose). The patient is prescribed antiemetics, pain relief, anticoagulant therapy, infusion therapy, gastric and intestinal motility stimulants. The patient starts drinking medical formula 24 hours after the end of surgical treatment. Postoperative physical activity - from 9.00 to 22.00 - walking for 10 minutes for every hour. The urinary catheter is removed 24 hours after the end of the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Tumor spread: cT2-4a cN0-3,
* cM0;
* Age: 18 - 80;
* Gender: men and women;
* ECOG: 0 - 1;
* Histologic type of tumor: Adenocarcinoma of any subtype;
* Degree of differentiation: G1 - G4;
* Tumor localization: cardiac region, stomach floor, stomach body, antrum, pylorus, and pyloric region of the stomach;
* Tumor spread: absence of tumor invasion into adjacent structures;
* No history of cancer in the last 5 years;
* No previous chemotherapy, surgery or radiation treatment for another cancer (except for neoadjuvant chemotherapy for gastric cancer);
* Absence of severe comorbidity restricting laparoscopic approach.

Exclusion Criteria:

* M1 (distant metastases);
* ECOG 2 - 4;
* Age over 80 and under 18;
* Presence of severe comorbidities, ASA> 3;
* Patient refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Investigation of the average number of lymph nodes removed during lymph node dissection using indocyanine green | 30 days after surgery

SECONDARY OUTCOMES:
Average number of metastatic ICG-positive lymph nodes | 30 days after surgery
Number of postoperative complications and complications associated with the introduction of ICG. | 90 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Available by request